CLINICAL TRIAL: NCT05970991
Title: Addressing Clinician Bias to Improve Equitable Implementation of Evidence-Based Practice-Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT)
Brief Title: Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT)
Acronym: VIBRANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Freda Liu, Assistant Professor: Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00016173; 1R34MH128386-01A1 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-08-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Implicit Bias
MeSH Terms: conditions — Bias, Implicit

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBC Controls (Active Comparator): Control group clinicians will complete the Brief Online Training (BOLT) for Measurement-Based Care (MBC) and consultation packages (4 online training modules supported by two 1-hour long, live post-training consultation sessions and expert-facilitated asynchronous online discussion board).
  Interventions: Behavioral: Brief Online Training (BOLT) for measurement-based care (MBC); Behavioral: Live Post-Training Consultation; Behavioral: Asynchronous Discussion Board
- MBC + VIBRANT (Experimental): Experimental condition clinicians will complete the same online training modules for MBC (BOLT) as the control group, but also complete the Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT) module (45 minutes). They will also receive two 1-hour long, live post-training consultation sessions and expert-facilitated asynchronous online discussion board.
  Interventions: Behavioral: Brief Online Training (BOLT) for measurement-based care (MBC); Behavioral: Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT); Behavioral: Live Post-Training Consultation; Behavioral: Asynchronous Discussion Board

INTERVENTIONS:
Behavioral: Brief Online Training (BOLT) for measurement-based care (MBC) — Brief Online Training (BOLT) for measurement-based care (MBC) is a series of 4 interactive, self-paced, online training modules that takes approximately 75 - 120 minutes to complete. Clinicians are trained on the core functions, procedures, and best practice approaches for delivering MBC in the school mental health setting. MBC is the systematic collection of patient-reported data to support collaborative clinical decision-making from intake to termination.
Behavioral: Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT) — The Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT) is a brief (45-minute), self-paced, interactive online training module designed to help school-based mental health clinicians understand and manage their implicit bias in clinical interactions.
  Arms: MBC + VIBRANT
Behavioral: Live Post-Training Consultation — Two 1-hour long small group consultation sessions with an expert consultant designed as additional opportunities to support knowledge elaboration and skills generalization.
Behavioral: Asynchronous Discussion Board — An expert facilitated online Discussion Board for additional opportunities of knowledge clarification, practice reinforcement, and community building to support implementation sustainment.

SUMMARY:
Healthcare providers' implicit bias has been identified as a contributor to longstanding health inequities via negative impacts on the patient-clinician relationship and biased delivery of high-quality evidence-based practices (EBP). The implementation of any EBP runs the risk of worsening existing health disparities due to inequitable access, delivery, or benefit of the intervention. Clinician bias can be a critical and unaddressed determinant of implementation for any EBP. Although some implicit bias interventions for healthcare providers are emerging, studies have rarely included mental health professionals. In a previously NIMH funded project, our research team iteratively developed a brief (~45 minutes), interactive online Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT) for school mental health clinicians with promising preliminary findings. The current study will test the effectiveness of VIBRANT-an implementation strategy for promoting equitable adoption, penetration, fidelity, and sustainment of EBPs. One highly learnable, efficient, and scalable EBP that is particularly well-suited for the education sector is Measurement-Base Care (MBC)-the systematic collection of patient-reported progress data to inform clinical decision-making. The proposed study aims to (1) evaluate VIBRANT's feasibility to promote equitable adoption, penetration, fidelity, and sustainment of MBC, with a validated, brief, interactive online training for MBC; (2) examine VIBRANT's impact on proximal mechanisms of change including clinicians' implicit bias as well as distal youth mental health outcomes (i.e., symptoms and functioning) with Black and Latinx youth, and (3) assess feasibility of research procedures for a future large-scale efficacy trial.

DETAILED DESCRIPTION:
Clinician bias constitutes a critical and unaddressed determinant of implementation for any Evidence-Based Practice (EBP). Implicit bias interferes with clinical decision-making and negatively impacts the clinician-patient relationship, leading ethnic/racial minoritized youth to receive suboptimal care resulting in disparate (worse) outcomes compared to their NHW peers. This is a preventable implementation gap (e.g., inequitable adoption, penetration, fidelity, sustainment) that substantially and unjustly limits the reach and public health impact of many of our most well-established EBPs in mental healthcare. This gap is particularly problematic in schools, where access to mental health services is significantly improved for ethnic minority youth, leading to more opportunities for disparate care quality. Despite the established knowledge base on implicit bias and bias reduction strategies, very little research has been done with mental health professionals; our team's previous work constitutes the first studies with mental health providers in the school setting. To address this gap in implicit bias intervention research and the lack of equity-focused implementation strategies, the investigators are conducting a pilot Hybrid Type 3 Effectiveness-Implementation Trial of a Virtual Implicit Bias Reduction and Neutralization Training (VIBRANT)-a highly efficient (~45 minutes), usable, and scalable intervention (interactive online training module) to address implicit bias among school mental health clinicians and support the equitable implementation of EBPs.

With previous NIMH funding, VIBRANT was iteratively developed for school mental health clinicians employing user-centered design principles. In a small proof-of-concept study (N = 12), school mental health clinicians found VIBRANT to be highly usable, appropriate, acceptable, and feasible to implement in their clinical practice. After completing the VIBRANT training, clinicians demonstrated notable improvements in implicit bias knowledge, and a downward trend in implicit bias (as measured by the Implicit Association Test) over 14 weeks. Moreover, clinicians with the greatest reductions in implicit bias also reported the strongest alliance with their youth patients. These results from our preliminary studies suggest that VIBRANT is an efficient and highly usable implementation strategy that holds promise for addressing clinician implicit bias to promote equitable implementation of other highly scalable evidence-based interventions.

Although VIBRANT is EBP-agnostic, it will be tested in the context of measurement-based care (MBC) implementation given (1) the high potential for MBC to optimize school mental health services, but currently inconsistent use in school mental health, and (2) MBC's vulnerability to inequitable delivery. Specifically, this study will evaluate the preliminary effectiveness of VIBRANT as an equity-focused implementation strategy for MBC. In addition to assessing VIBRANT's impact on equitable MBC adoption, penetration, fidelity, and sustainment within and between clinician caseloads, the investigators will also examine impact on proximal mechanisms of change (clinician implicit bias, therapeutic alliance) and distal youth clinical and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for each of the subjects participating in the study as follows:

1. Participating clinicians must…

   1. Provide school-based mental health services in middle and high school settings for at least 50% of their clinical deployment.
   2. Provide on-going 1:1 mental health services to students (e.g., not assessment only).
   3. Have a caseload (who is receiving on-going care) that consists of at least 20% of Black or Latinx students.
2. Participating youths must…

   1. Identify as Black/African American or/and Hispanic/Latina/Latino/Latinx
   2. be entering into ongoing treatment with a participating clinician in the school mental health setting
3. Participating caregivers must… a. be a primary caregiver to the youth who can answer questions about the youth's daily behaviors and emotional well-being

Exclusion Criteria:

Exclusion criteria for each of the subjects participating:

1. School-based mental health clinicians

   1. Clinician who previously participated in a measurement-based care (MBC) related study with our team and have already been exposed to our online MBC training.
   2. Clinicians who have participated in a previous study related to VIBRANT.
2. Black & Latinx youth

   1. Youths with a developmental or learning disability that would interfere with their ability to accurately give informed consent or assent and reliable completion of study assessments.
   2. Youths who do not speak English or Spanish
3. Caregivers

   1. Caregivers who do not reside with the youth or would otherwise have adequate daily contact to report on the youth's typical behaviors and/or emotional well-being.
   2. Caregiver who do not speak English or Spanish

Ages: 11 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Adoption of Measurement-Based Care (MBC) strategies | 4-month (follow-up 2)
  Clinicians will complete weekly caseload service logs, that document whether each of the 3 core MBC practices (i.e., measure administration, clinician reviewing results, discussing results with patient to support collaborative treatment planning) were used with each identified patient in their caseload. MBC adoption (client level) will be a binary measure for each youth on the clinicians' caseload-evidence of any MBC practice will be considered adoption. This is a longitudinal outcome that will be collected on a weekly basis to allow for the observation of growth over time.
Penetration or saturation of Measurement-Based Care (MBC) strategies use | 4-month (follow-up 2)
  Clinicians will complete weekly caseload service logs, that document whether each of the 3 core MBC practices (i.e., measure administration, clinician reviewing results, discussing results with patient to support collaborative treatment planning) were used with each identified patient on their caseload. MBC penetration will be derived from dividing the number of youths on the clinician's caseload who is receiving any MBC practices by the total number of youths on the caseload, which should yield a percentage score.
Sustainment of Measurement-Based Care (MBC) strategies use | 4-month (follow-up 2)
  Clinicians will complete weekly caseload service logs, that document whether each of the 3 core MBC practices (i.e., measure administration, clinician reviewing results, discussing results with patient to support collaborative treatment planning) were use with each identified patient on their caseload. MBC sustainment will be indicated by the change in MBC penetration at 1 months post-training (Follow-Up 1) and 3 months post-training (Follow-Up 2).
Fidelity of Measurement-Based Care (MBC) Strategies use | 4-month (follow-up 2)
  Clinicians will complete weekly caseload service logs, that document whether each of the 3 core MBC practices (i.e., measure administration, clinician reviewing results, discussing results with patient to support collaborative treatment planning) were used with each identified patient on their caseload. Fidelity will be measured by percentage of a clinician's caseload with whom all 3 MBC core components were reported on their caseload service logs.
Change in Clinician's Implicit Association Test (IAT) Scores | 0-months (Pre-training), 1-month (post-training), 2-month follow-up 1, and 4-month (follow-up 2)
  The Implicit Association Test (IAT), the most well-established measure of implicit racial attitudes with over 20 years of empirical support, is a computer-based reaction time task that measures the relative strength of association between pairings of two groups with two evaluative attributes (e.g., White-good and Black-bad vs White-bad and Black-good). The difference in reaction time between the two pairings would reveal the respondent's relative bias. Clinicians will complete 4 distinct IATs (via the online surveys) at each data collection timepoint. The IATs will measure (1) implicit prejudice toward Black (2) and Latinx youth (both in comparison to White youth), (3) implicit stereotyping of Black youth as aggressive compared to White youth (peaceful), and (4) implicit stereotyping of Latinx youth associated with academic failure and White youth with academic success.
Change in Clinician and Youth Working Alliance Inventory--Short Form scores | 1-month (post-training), 4-month (follow-up 2)
  Working Alliance Inventory--Short Form is a 12-item clinician- and patient-report rating scale of the therapeutic relationship with items that capture agreement on the goals and tasks of therapy as well as the therapeutic bond. It has been validated for use with youth 11-18 years old, demonstrating excellent internal consistency (α = 0.93 to 0.96) for both youth and clinician rating forms, and evidencing a single factor structure.
Change in Strengths and Difficulties Questionnaire (SDQ) youth and caregiver report scores | 1-month (post-training), 4-month (follow-up 2)
  The Strengths and Difficulties Questionnaire (SDQ) is a 25-item self- and informant-reported symptom questionnaire that has been validated for use with youths ages 4-18 (self-report for 11-18+) with 5 subscales (emotional distress, conduct problems, attention, peer relationships, prosocial behaviors). Internal consistency for these subscales is adequate, ranging from α = .78 to .82. An additional 5 items comprise an "impact scale" that assesses the degree to which youth's symptoms interfere with different domains of functioning. The impact and prosocial subscale scores will serve as our measures of functional impairment. The SDQ has demonstrated strong psychometrics in large-scale studies with US and international samples and has been shown to be sensitive to treatment change. Spanish versions have been validated with evidence of similar factor structure, measurement invariance, and adequate internal consistency for both youth and parent report, α = .71 to .75.

CONTACTS AND LOCATIONS:
Overall Officials: Freda Liu, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatty GB. Subdural haematoma: an evaluation of treatment methods. J Indian Med Assoc. 1996 Jan;94(1):7-10. PMID 8776032
- [Background] Sampson BK, Doran KA. Health needs of coronary artery bypass graft surgery patients at discharge. Dimens Crit Care Nurs. 1998 May-Jun;17(3):158-64; quiz 165-8. doi: 10.1097/00003465-199805000-00009. PMID 9633346
- [Background] Garcia-Segura LM, Rodriguez JR, Torres-Aleman I. Localization of the insulin-like growth factor I receptor in the cerebellum and hypothalamus of adult rats: an electron microscopic study. J Neurocytol. 1997 Jul;26(7):479-90. doi: 10.1023/a:1018581407804. PMID 9306246